CLINICAL TRIAL: NCT00440765
Title: A Post Authorization Study, Designed to Learn More About the Safety and Efficacy of the Use of VELCADE (Bortezomib) in the Netherlands
Brief Title: VALEO: A Post Authorization Study, Designed to Learn More About the Safety and Effectiveness of the Use of Bortezomib in the Netherlands
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR003469; 26866138MMY4001
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Multiple Myeloma; Hematological Neoplasms
Keywords: Multiple Myeloma; hematological Neoplasms; chemotherapy; efficacy; safety; bortezomib; proteasome inhibitor
MeSH Terms: conditions — Multiple Myeloma; Hematologic Neoplasms | interventions — Bortezomib

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 001: bortezomib dose as determined (observational study) by treating physician
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — dose as determined (observational study) by treating physician

SUMMARY:
The main purpose of this study is to evaluate safety and effectiveness of the treatment of multiple myeloma with bortezomib in daily practice in the Netherlands.

DETAILED DESCRIPTION:
Bortezomib has become commercially available in the European Union in May 2004 for the third line treatment of patients with multiple myeloma. The registration was based on two phase II studies while more research was ongoing. Some experience was already gained with the use of this product in the Netherlands by means of a compassionate use program before the initial registration. However, the data available from the use of bortezomib in daily clinical practice is limited. Therefore, there is a need to closely study the use of bortezomib in daily clinical practice. During the course of the study, the registration of bortezomib was extended. In April 2005, bortezomib was registered for second line treatment of multiple myeloma. Consequently, safety and effectiveness data from patients in this line of treatment could be collected in this project as well (arm A). Data of a large phase 3 trial showed that response rates differ between patients treated for multiple myeloma in the second line and patients treated in the third line. Therefore the protocol was amended to compare the response rates in two arms, dependent on the number of previous treatment lines for multiple myeloma: The protocol was also amended to determine the time to progression and response rate in both patients who received thalidomide earlier versus patients who didn't (arm B). ARM A: Patients with relapsed multiple myeloma who have received not more than 1 previous line of treatment and show progression on that therapy; ARM B: Patients with relapsed or refractory multiple myeloma who have received at least 2 prior lines of treatment and show progression on most recent therapy. This project is a 'post authorization study (PAS)'. This means that only routinely available medical data is collected, with the patients' permission, and no additional interventions or diagnostic procedures should be done specifically for this study. Because the study is observational, dosage, administration and duration of treatment is at discretion of treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients have to sign a statement that they agree with collection of their clinical data for this project
* the patient is eligible, in the investigator's opinion, based on the criteria in the summary of product characteristics for bortezomib

Exclusion Criteria:

* If patients meet the eligibility criteria, there are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Myeloma patients treated with bortezomib in second or later line of therapy
Sampling Method: Non-Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2004-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Response to treatment; determination of response, duration of response, determination of relapse/progression | no timepoints are defined, as this is an observational study; data will be collected until three years after last bortezomib administration.

SECONDARY OUTCOMES:
bortezomib treatment schedule used | each cycle
combination therapies for multiple myeloma | from start of bortezomib treatment up to 30 days after last bortezomib administration
adverse events | from start of bortezomib treatment up to 30 days after last bortezomib administration
overall survival | from end of bortezomib treatment up to 3 years after last bortezomib administration

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag B.V. Clinical Trial, Study Director — Janssen-Cilag B.V.
Locations (44):
- Netherlands (44):
  - 's-Hertogenbosch
  - Alkmaar
  - Amersfoort
  - Amstelveen
  - Amsterdam-Zuidoost
  - Apeldoorn
  - Bergen op Zoom
  - Blaricum
  - Breda
  - Capelle Aan Den Ijss
  - Delfzijl
  - Deventer
  - Dirksland
  - Doetinchem
  - Dordrecht
  - Drachten
  - Ede Gld
  - Eindhoven
  - Flushing
  - Geldrop
  - Goes
  - Gouda
  - Groningen
  - Hardenberg
  - Heerenveen
  - Hoofddorp
  - Hoogeveen
  - Leiden
  - Maastricht
  - Nieuwegein
  - Nijmegen
  - Oss
  - Roosendaal
  - Rotterdam
  - Schiedam
  - Terneuzen
  - The Hague
  - Tilburg
  - Utrecht
  - Veghel
  - Veldhoven
  - Woerden
  - Zaandam
  - Zutphen